CLINICAL TRIAL: NCT03279666
Title: A Randomized Controlled Study: Patients' With or Without Tenaculum Placement and Intracervical Blockage/or Not During Colposcopic Biopsy
Brief Title: Biopsy Size and Pain Perception During Colposcopic Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2017/47
Record Dates: First submitted 2017-08-16; First posted 2017-09-12 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Pain Uterus; Tenaculum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tenaculum with intracervical blockage (Active Comparator)
  Interventions: Other: Tenaculum replacement
- No tenaculum with intracercical blockage (No Intervention)
- Tenaculum without intracervical blockage (Active Comparator)
  Interventions: Other: Tenaculum replacement
- No Tenaculum without intracervical blockage (No Intervention)

INTERVENTIONS:
Other: Tenaculum replacement — Tenaculum replacement during colposcopic biopsy
  Arms: Tenaculum without intracervical blockage; tenaculum with intracervical blockage

SUMMARY:
The investigators will investigate patients pain and biopsy size during colposcopic biopsy. The investigators will use tenaculum randomized patient with or without intracervical blockage.

DETAILED DESCRIPTION:
The study was designed four arms. The investigators will perform colposcopy because of various causes. The first arm is used tenaculum and performed intracervical blockage. The second arm is not used tenaculum and performed intracervical blockage. The third arm is used tenaculum and not performed intracervical blockage. The fourth arm is not used tenaculum and not performed intracervical blockage and then we will study patients pain and biopsy size during colposcopic biopsy. Pain reduce and biopsy size are very important for patient and diagnose of the cervix cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 year-old women who had colposcopic biopsy

Exclusion Criteria:

* Had orthopedical problems
* Analgesic allergy
* Have previous cone biopsy
* Analgesic use until six hours before colposcopy
* Advanced cervicovaginal atrophy
* Linear Visual Analog Score for pain is used

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Patients' Biopsy Sizes | 6 months
  Are patients' biopsy sizes associate with tenaculum. Milimeter will be used for biopsy size.
Patients' Biopsy Sizes | 6 months
  Are patients' biopsy sizes associate with analgesic. Milimeter will be used for biopsy size.

SECONDARY OUTCOMES:
Patients' pain perceptions | 6 months analgesic
  Are patients' pain perceptions associate with analgesic. Linear Visual Analog Scale will be used for pain perception.
Patients' pain perceptions | 6 months
  Are patients' pain perceptions associate with teanaculum. Linear Visual Analog Scale will be used for pain perception.

CONTACTS AND LOCATIONS:
Locations (1):
- Cihan Comba, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Comba C, Demirayak G, Erdogan SV, Karaca I, Demir O, Guler O, Ozdemir IA. Comparison of pain and proper sample status according to usage of tenaculum and analgesia: a randomized clinical trial. Obstet Gynecol Sci. 2020 Jul;63(4):506-513. doi: 10.5468/ogs.19185. Epub 2020 Jun 19. PMID 32550738